CLINICAL TRIAL: NCT04863703
Title: Improvement of Portal Hypertension During Viral Suppression in Patients With Hepatitis Delta (IMPHROVE-D)
Acronym: IMPHROVE-D
Status: Active, not recruiting | Type: Observational
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Maasoumy, Benjamin PD Dr, PD Dr. med. Benjamin Maasoumy, Hannover Medical School
Other Study IDs: 9644_BO_S_2021
Record Dates: First submitted 2021-04-13; First posted 2021-04-28 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-03

CONDITIONS: Hepatitis D; Hepatitis B; Portal Hypertension; Liver Cirrhosis
Keywords: Portal hypertension, Liver cirrhosis, Bulevirtide, Hepatitis D, Hepatitis B
MeSH Terms: conditions — Hepatitis D; Hepatitis B; Hypertension, Portal; Liver Cirrhosis | interventions — bulevirtide

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- One group with HBV/HDV coinfection: Measurement of HVPG before antiviral treatment of HBV/HDV coinfection and one year after treatment initiation with Bulevirtide. Administration of Bulevirtide and HVPG measurement is independent from this study.
  Interventions: Drug: Bulevirtide

INTERVENTIONS:
Drug: Bulevirtide — Patients with liver cirrhosis and HBV/HDV coinfection receive Bulevirtide as an antiviral therapy irrespective of the study, this study is observational.

SUMMARY:
Portal hypertension (PH) is one of the key drivers of clinical deteoration in patients with liver cirrhosis. It has been demonstrated that antiviral therapy in patients with chronic hepatitis C infection leads to a decrease of PH and is associated with an improved outcome. Recently, Bulevirtide was approved for the treatment of patients coinfected with hepatitis B (HBV) and chronic hepatitis delta (HDV) infection, which helps to achieve viral supression in these patients. This study investigates the potential effects of viral supression on PH in patients with chronic HBV/HDV infection and liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HBV/HDV Coinfection
* suspected or diagnosed liver cirrhosis, indication for hepatovenous pressure gradient (HVPG) measurement or liver cirrhosis and HVPG measurement conducted in the past 12 months (conducted prior to antiviral treatment)
* indication for antiviral treatment with Bulevirtide
* age >18years
* Must be willing to participate in the study and provide written informed consent

Exclusion Criteria:

* patient rejects study participation
* no conducted or no indication for HVPG measurement
* age <18years

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study populations consists out of patients with HBV/HDV coinfection, diagnosed or suspected liver cirrhosis. All patients must have a medical indication for HVPG measurement or had a HVPG measurement within the last 12 months.
Sampling Method: Probability Sample
Enrollment: 11 (Estimated)
Dates: Start 2021-05-07 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change the degree of portal hypertension after inducing viral suppression via antiviral treatment with Bulevirtide | Measurement before antiviral treatment (baseline) and one year after inducing viral suppression with Bulevirtide.
  Change of hepatovenous pressure gradient (HVPG) in mmHg underviral suppression with Bulevirtide in patients with HBV/HDV coinfection and liver cirrhosis. HVPG measurement will be assessed via transjugular HVPG measurement.

SECONDARY OUTCOMES:
Change of Quality of life under viral suppression with Bulevirtide | Measurement before Bulevirtide intake (baseline) and one year after establishing antiviral treatment.
  Change of Quality of life is assessed via SF-36 questionnaire.
Change in minimal hepatic encephalopathy (HE) status under viral suppression | Measurement before antiviral treatment (baseline) and one year after inducing viral suppression with Bulevirtide.
  Change in minimal HE status is evaluated via PSE-testing, critical flicker frequency and animal naming test.
Change of nutritional status under viral suppression with Bulevirtide | Measurement before antiviral treatment (baseline) and one year after inducing viral suppression with Bulevirtide.
  Change of nutritional status will be evaluated via repeated measurement of BMI (in kg/m2), arm circumference and triceps skin fold thickness.
Change of physical ability under viral suppression with Bulevirtide | Measurement before antiviral treatment (baseline) and one year after inducing viral suppression with Bulevirtide.
  Change of physical ability is assessed via liver-frailty Index.
Change of the inflammatory profile under viral suppression with Bulevirtide | Measurement before antiviral treatment (baseline) and one year after inducing viral suppression with Bulevirtide.
  Change of the inflammatory profile will be assessed through Cytokines using Bio-Plex Pro Human Cytokine Screening Panel, 48-Plex, Bio-Rad, Olink Target 96 Inflammation and Olink Proteomics.
Change in liver stiffness under viral suppression with Bulevirtide | Measurement before Bulevirtide intake (baseline) and one year after establishing antiviral treatment with Bulevirtide.
  Change in liver stiffness will be assessed via transient elastography.
Clinical endpoints under viral suppression with Bulevirtide | Measurement before antiviral treatment (baseline) and one year after inducing viral suppression with Bulevirtide.
  Assessed clinical endpoints are: Resolution of esophageal varices and incidence of esophageal bleeding, hepatic encephalopathy or ascites.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Maasoumy, MD, Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided